CLINICAL TRIAL: NCT00340132
Title: Cross-Sectional and Longitudinal Studies of 'Pre-Diabetes'
Brief Title: Cross-Sectional and Longitudinal Studies of "Pre-Diabetes" in the Pima Indians
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 9999820136; OH82-DK-0136
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-17

CONDITIONS: Weight Gain; Overweight; Insulin Resistance; Obesity; Diabetes Mellitus, Type 2
Keywords: Insulin Sensitivity; Insulin Secretion; Glucose Tolerance; Adipose Tissue; Preadipocytes; Natural History
MeSH Terms: conditions — Weight Gain; Overweight; Insulin Resistance; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult volunteers: Volunteers aged 18-55 who are healthy as determined by medical history, physical examination, and laboratory tests

SUMMARY:
Insulin resistance and a defect in early insulin secretion are risk factors for the development of type 2 diabetes mellitus. A recent longitudinal analysis which tracked the development of diabetes demonstrated that both insulin action and early insulin secretion deteriorate as individuals progress from normal to impaired glucose tolerance and then to diabetes. These results suggest that both inherent (apparent in normal glucose tolerant subjects who progress to diabetes and likely to have a genetic basis) and acquired (evident as individuals progress from NGT to IGT to diabetes and possibly environmental in origin) defects in insulin action and secretion contribute to the pathogenesis of type 2 diabetes. To identify the genetic and environmental determinants of diabetes we are continuing to determine: (1) if there are genes that segregate with metabolic risk factors for diabetes which might therefore be genetic markers for type 2 diabetes and (2) the mechanisms mediating genetic and environmental determinants of insulin resistance and impaired insulin secretion.

<TAB>

Volunteers for this study will be admitted to the clinical research ward where they will undergo several tests to determine body composition, oral and intravenous glucose tolerance and in vivo insulin action. In addition, in selected subjects, adipose and/or skeletal muscle tissue will be obtained by percutaneous biopsy for in vitro studies of gene expression and insulin action in these tissues. A transformed lymphocyte cell line will be established for each subject as a permanent source of DNA for genetic studies. Genetic markers for type 2 diabetes and insulin resistance will be sought by typing each individual at positional and functional candidate loci in the hopes of finding an association between these loci and obesity, insulin secretion, insulin resistance and/or type 2 diabetes.

DETAILED DESCRIPTION:
Insulin resistance and a defect in early insulin secretion are risk factors for the development of type 2 diabetes mellitus. A recent longitudinal analysis which tracked the development of diabetes demonstrated that both insulin action and early insulin secretion deteriorate as individuals progress from normal to impaired glucose tolerance and then to diabetes. These results suggest that both inherent (apparent in normal glucose tolerant subjects who progress to diabetes and likely to have a genetic basis) and acquired (evident as individuals progress from NGT to IGT to diabetes and possibly environmental in origin) defects in insulin action and secretion contribute to the pathogenesis of type 2 diabetes. To identify the genetic and environmental determinants of diabetes we are continuing to determine: (1) if there are genes that segregate with metabolic risk factors for diabetes which might therefore be genetic markers for type 2 diabetes and (2) the mechanisms mediating genetic and environmental determinants of insulin resistance and impaired insulin secretion.

<TAB>

Volunteers for this study will be admitted to the clinical research ward where they will undergo several tests to determine body composition, oral and intravenous glucose tolerance and in vivo insulin action. In addition, in selected subjects, adipose and/or skeletal muscle tissue will be obtained by percutaneous biopsy for in vitro studies of gene expression and insulin action in these tissues. A transformed lymphocyte cell line will be established for each subject as a permanent source of DNA for genetic studies. Genetic markers for type 2 diabetes and insulin resistance will be sought by typing each individual at positional and functional candidate loci in the hopes of finding an association between these loci and obesity, insulin secretion, insulin resistance and/or type 2 diabetes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects from all racial and ethnic backgrounds will be invited to participate if they are:

* Ages: 18-55 years old (up to 2200 participants)
* Gender: male or female

EXCLUSION CRITERIA:

Subjects will be excluded who are:

* Taking medication for a chronic illness.
* Have any acute or chronic diseases or conditions not specifically mentioned that in the opinion of the provider may interfere with the study or decrease safety for participation will be considered exclusionary.
* Women who currently pregnant or breastfeeding.
* Positive for drug and/or nicotine use.

All medications and alcohol consumption are to be stopped for two weeks prior to admission. A urine drug-screening test for drugs such as narcotics, marijuana, and barbiturates will be performed on everyone to exclude from the study people whose urine show active or recent drug use. A positive drug test could confound the results of the study in an unpredictable manner. The results of this test will become a part of the patient s medical records and may be released if requested (please see page 6 of the consent for details regarding medical records release).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample from eligible participants from greater Phoenix metropolitan area@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 1759 (Actual)
Dates: Start 1983-01-01 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance via oral glucose tolerance test (OGTT) | Baseline, and after 180 minutes on day 4
  Measured via OGTT after ingestion of 75 grams of glucose over 2 minutes
Glucose tolerance via intravenous glucose tolerance test (IVGTT) | Baseline and after 10 minutes on day 5
  Measured via IVGTT after administration of a glucose bolus (25 g as a 50% solution injected over 3 minutes)
Basal endogenous glucose production | Baseline, and after 100 minutes on day 10
  Assessed using deuterium (D-6,6 2H) glucose as a tracer, infused as a 10 mL bolus followed by 0.150 mL/min for a total of 350 minutes
24-hour metabolic rate | Baseline and after 23.5 hours on day 7
  Assessed from the rates of caloric expenditure and substrate utilization while in the human respiratory chamber for 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Votruba, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Mitchell CM, Stinson EJ, Chang DC, Krakoff J. A mixed meal tolerance test predicts onset of type 2 diabetes in Southwestern Indigenous adults. Nutr Diabetes. 2024 Jul 10;14(1):50. doi: 10.1038/s41387-024-00269-3. PMID 38987291
- [Derived] Aydin BN, Stinson EJ, Cabeza De Baca T, Ando T, Travis KT, Piaggi P, Krakoff J, Chang DC. Investigation of seasonality of human spontaneous physical activity and energy expenditure in respiratory chamber in Phoenix, Arizona. Eur J Clin Nutr. 2024 Jan;78(1):27-33. doi: 10.1038/s41430-023-01347-y. Epub 2023 Oct 13. PMID 37833567
- [Derived] Stinson EJ, Mitchell CM, Looker HC, Krakoff J, Chang DC. Higher glucose and insulin responses to a mixed meal are associated with increased risk of diabetic retinopathy in Indigenous Americans. J Endocrinol Invest. 2024 Mar;47(3):699-707. doi: 10.1007/s40618-023-02187-0. Epub 2023 Sep 9. PMID 37684485
- [Derived] Basolo A, Ando T, Chang DC, Hollstein T, Krakoff J, Piaggi P, Votruba S. Reduced Albumin Concentration Predicts Weight Gain and Higher Ad Libitum Energy Intake in Humans. Front Endocrinol (Lausanne). 2021 Mar 11;12:642568. doi: 10.3389/fendo.2021.642568. eCollection 2021. PMID 33776937
- [Derived] Shah MH, Piaggi P, Looker HC, Paddock E, Krakoff J, Chang DC. Lower insulin clearance is associated with increased risk of type 2 diabetes in Native Americans. Diabetologia. 2021 Apr;64(4):914-922. doi: 10.1007/s00125-020-05348-5. Epub 2021 Jan 6. PMID 33404681
- [Derived] Piaggi P, Koroglu C, Nair AK, Sutherland J, Muller YL, Kumar P, Hsueh WC, Kobes S, Shuldiner AR, Kim HI, Gosalia N, Van Hout CV, Jones M, Knowler WC, Krakoff J, Hanson RL, Bogardus C, Baier LJ. Exome Sequencing Identifies A Nonsense Variant in DAO Associated With Reduced Energy Expenditure in American Indians. J Clin Endocrinol Metab. 2020 Nov 1;105(11):e3989-4000. doi: 10.1210/clinem/dgaa548. PMID 32818236
- [Derived] Heinitz S, Gebhardt C, Piaggi P, Kruger J, Heyne H, Weiner J, Heiker JT, Stumvoll M, Bluher M, Baier L, Rudich A, Kovacs P, Tonjes A. Atg7 Knockdown Reduces Chemerin Secretion in Murine Adipocytes. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5715-5728. doi: 10.1210/jc.2018-01980. PMID 31225870
- [Derived] Heinitz S, Basolo A, Piomelli D, Krakoff J, Piaggi P. Endocannabinoid Anandamide Mediates the Effect of Skeletal Muscle Sphingomyelins on Human Energy Expenditure. J Clin Endocrinol Metab. 2018 Oct 1;103(10):3757-3766. doi: 10.1210/jc.2018-00780. PMID 30113648
- [Derived] Heinitz S, Piaggi P, Yang S, Bonfiglio S, Steel J, Krakoff J, Votruba SB. Response of skeletal muscle UCP2-expression during metabolic adaptation to caloric restriction. Int J Obes (Lond). 2018 Jun;42(5):974-984. doi: 10.1038/s41366-018-0085-2. Epub 2018 May 17. PMID 29777235
- [Derived] Heinitz S, Basolo A, Piaggi P, Piomelli D, Jumpertz von Schwartzenberg R, Krakoff J. Peripheral Endocannabinoids Associated With Energy Expenditure in Native Americans of Southwestern Heritage. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1077-1087. doi: 10.1210/jc.2017-02257. PMID 29300902
- [Derived] Piaggi P, Masindova I, Muller YL, Mercader J, Wiessner GB, Chen P; SIGMA Type 2 Diabetes Consortium; Kobes S, Hsueh WC, Mongalo M, Knowler WC, Krakoff J, Hanson RL, Bogardus C, Baier LJ. A Genome-Wide Association Study Using a Custom Genotyping Array Identifies Variants in GPR158 Associated With Reduced Energy Expenditure in American Indians. Diabetes. 2017 Aug;66(8):2284-2295. doi: 10.2337/db16-1565. Epub 2017 May 5. PMID 28476931
- [Derived] Hohenadel MG, Baier LJ, Piaggi P, Muller YL, Hanson RL, Krakoff J, Thearle MS. The impact of genetic variants on BMI increase during childhood versus adulthood. Int J Obes (Lond). 2016 Aug;40(8):1301-9. doi: 10.1038/ijo.2016.53. Epub 2016 Apr 14. PMID 27076275
- [Derived] Piaggi P, Thearle MS, Bogardus C, Krakoff J. Fasting hyperglycemia predicts lower rates of weight gain by increased energy expenditure and fat oxidation rate. J Clin Endocrinol Metab. 2015 Mar;100(3):1078-87. doi: 10.1210/jc.2014-3582. Epub 2015 Jan 5. PMID 25559400
- [Derived] Piaggi P, Krakoff J, Bogardus C, Thearle MS. Lower "awake and fed thermogenesis" predicts future weight gain in subjects with abdominal adiposity. Diabetes. 2013 Dec;62(12):4043-51. doi: 10.2337/db13-0785. Epub 2013 Aug 23. PMID 23974925